CLINICAL TRIAL: NCT00869921
Title: Attain StarFix® Model 4195 Left Ventricular Lead Chronic Performance Post Approval Study
Brief Title: Model 4195 Left Ventricular (LV) Lead Chronic Performance Study
Status: Completed | Type: Observational
Sponsor: Medtronic (Industry)
Responsible Party: Sponsor
Other Study IDs: 4195 Chronic Performance
Record Dates: First submitted 2009-03-25; First posted 2009-03-26 (Estimated); Last update posted 2018-09-13 (Actual); Status verified 2018-09

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Evaluate long-term performance of the 4195 LV Lead. This evaluation is based on the number of lead-related complications occuring during the study compared to the number of leads enrolled in the study. The leads will be followed for 5 years after implant. This study is required by FDA as a condition of approval of the Model 4195 LV Lead and is integrated within Medtronic's post-market surveillance platform.

DETAILED DESCRIPTION:
Model 4195 LV lead complication-free survivability will be summarized.

ELIGIBILITY:
Patients who meet all of the following inclusion criteria and do not meet any of the following exclusion criteria are eligible for enrollment.

Inclusion Criteria

* Patient or legally authorized representative provides written authorization and/or consent per institution and geographical requirements
* Patient has or is intended to receive an Attain StarFix Model 4195 LV lead
* Patient within 30 day post implant enrollment window

Exclusion Criteria

* Patient who is, or is expected to be inaccessible for follow-up
* Patient with exclusion criteria required by local law
* Patient is currently enrolled in or plans to enroll in any concurrent drug and/or device study that may confound results

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients implanted with a 4195 LV Lead within the past 30 days. All patients must meet Inclusion criteria and none of the Exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 1322 (Actual)
Dates: Start 2009-03; Primary Completion 2018-04-03 (Actual); Study Completion 2018-04-03 (Actual)

PRIMARY OUTCOMES:
Lead-related complication rate. | Implant to 5 years post-implant.

SECONDARY OUTCOMES:
Types of Model 4195 lead-related events | 5 years post implant

CONTACTS AND LOCATIONS:
Overall Officials: 4195 LV Lead Chronic Performance Study Team, Study Chair — Medtronic
Locations (67):
- United States (62):
  - Anchorage, Alaska
  - Phoenix, Arizona
  - Scottsdale, Arizona
  - Chula Vista, California
  - Redding, California
  - Salinas, California
  - Stanford, California
  - Torrance, California
  - Colorado Springs, Colorado
  - New Haven, Connecticut
  - Bradenton, Florida
  - Clearwater, Florida
  - Jacksonville, Florida
  - Melbourne, Florida
  - Albany, Georgia
  - Marietta, Georgia
  - Indianapolis, Indiana
  - Newburgh, Indiana
  - Des Moines, Iowa
  - Kansas City, Kansas
  - Edgewood, Kentucky
  - Louisville, Kentucky
  - Baton Rouge, Louisiana
  - Covington, Louisiana
  - Salisbury, Maryland
  - Silver Spring, Maryland
  - Takoma Park, Maryland
  - Boston, Massachusetts
  - Grand Blanc, Michigan
  - Marquette, Michigan
  - Robbinsdale, Minnesota
  - Rochester, Minnesota
  - Saint Louis Park, Minnesota
  - Columbia, Missouri
  - Kansas City, Missouri
  - Henderson, Nevada
  - West Orange, New Jersey
  - Albuquerque, New Mexico
  - New York, New York
  - Durham, North Carolina
  - Fargo, North Dakota
  - Cincinnati, Ohio
  - Cleveland, Ohio
  - Columbus, Ohio
  - Toledo, Ohio
  - Portland, Oregon
  - Lancaster, Pennsylvania
  - Germantown, Tennessee
  - Kingsport, Tennessee
  - Nashville, Tennessee
  - Austin, Texas
  - Dallas, Texas
  - Fort Worth, Texas
  - Houston, Texas
  - Plano, Texas
  - San Antonio, Texas
  - Burlington, Vermont
  - Falls Church, Virginia
  - Olympia, Washington
  - Spokane, Washington
  - Madison, Wisconsin
  - Milwaukee, Wisconsin
- Canada (4):
  - Calgary, Alberta
  - Kingston, Ontario
  - Ottawa, Ontario
  - Québec, Quebec
- Middlesbrough, United Kingdom